CLINICAL TRIAL: NCT06546930
Title: Optimizing Diabetes Technology Use for Latinx Youth Through DREAM (Device Use Reimagined Through Education And Mentorship) Virtual Peer Groups [Study-wide] - DREAM Intervention
Brief Title: Device Use Reimagined Through Education And Mentorship
Acronym: DREAM
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, San Francisco (Other)
Collaborators: Children's Hospital Los Angeles (Other); University of California, Davis (Other); National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 24-41906; 5R01DK135000 (NIH)
Record Dates: First submitted 2024-08-02; First posted 2024-08-09 (Actual); Last update posted 2025-10-15 (Actual); Status verified 2025-10

CONDITIONS: Diabetes Mellitus, Type 1
Keywords: T1D; Diabetes; Diabetes Mellitus; Type 1
MeSH Terms: conditions — Diabetes Mellitus, Type 1; Diabetes Mellitus

STUDY DESIGN:
Intervention Model Description: Intervention group (will receive VPG curriculum) versus comparator group (not enrolled)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Experimental): Virtual peer groups (VPGs)
  Six different VPGs topics will be offered. Each VPG topic will be presented separately to youth and caregivers, in Spanish and English. Frequency of scheduling for each VPG will vary on a month-to-month basis depending on the distribution of current enrollees who have not yet discussed that topic and the availability of the relevant facilitators.
  In-Person Events
  Optional in-person events may be offered quarterly during the 6-12 month study participation period.
  Interventions: Behavioral: DREAM intervention
- Comparator Group (No Intervention): An equal number of eligible non-enrolled patients at each site will be selected and matched to the enrolled cohort based on age, language, HbA1c, insurance type, and diabetes technology use at a population level.

INTERVENTIONS:
Behavioral: DREAM intervention — Virtual Peer Groups (VPGs)
  Participants will have multiple opportunities to attend a VPG on a specific topic during their 6-12 month participation period. The VPG topics will include the following:
  * Diabetes technology - basics or advanced use (audience-dependent)
  * Family relationships and diabetes
  * Diabetes in real life - school, work, social gatherings, travel
  * Wellbeing and support when living with diabetes
  * Working with your diabetes care team - who to call for what
  * Eating and activity - what's different with T1D?
  In-Person Events will be held quarterly to facilitate participant interaction and community-building. These gatherings will feature ice-breaker activities, refreshments, and hands-on learning opportunities, including the chance to interact with specific diabetes devices and engage with healthcare professionals and representatives from diabetes technology companies.
  Arms: Intervention

SUMMARY:
Diabetes technology, such as insulin pumps and continuous glucose monitoring devices, can help improve glucose control for people with type 1 diabetes (T1D), which keeps them at lower risk for diabetes complications, but many Latinx adolescents, who make up the largest marginalized ethnic group of youth with T1D in California, use these devices less often and have less optimal glucose control compared to White youth. In phase 1 of this project, we worked directly with Latinx youth, their families, and diabetes care team members in California to develop DREAM, Device use Reimagined through Education And Mentorship, a virtual peer group (VPG) intervention that will encourage and support the use of diabetes devices in Latinx adolescents with T1D. The goals for phase 2 (intervention) of this project are to evaluate the feasibility and acceptability of the stakeholder-informed VPG intervention, and evaluate clinical and person-centered outcomes.

DETAILED DESCRIPTION:
This multi-site project has two phases: phase 1 involved stakeholders focus groups to assess barriers and facilitators to diabetes technology and the creation of advisory councils. Feedback was obtained and used to develop phase 2, the single arm trial. A virtual peer group curriculum is being refined and will be implemented. The aims of this project are: (1) Partner with stakeholders to design a virtual peer group (VPG) intervention to promote the initiation and continued use of diabetes technology among Latinx adolescents with T1D. (2) Evaluate the feasibility and acceptability of DREAM VPGs in a pragmatic, single arm trial. (3) Assess the effects of DREAM VPGs on clinical and person-centered outcomes.

Our DREAM intervention will:

* Build trust/rapport and "relational connections" between participants
* Empower participants to be advocates in their/their adolescents' diabetes care
* Provide tools/knowledge to navigate healthcare and diabetes technology systems
* Increase knowledge, confidence, and interest in using diabetes technology
* Create a culturally sensitive/inclusive VPG toolkit that will be scalable, feasible, and sustainable in broader clinical contexts if found to be beneficial

The DREAM project's findings will inform future efforts to improve diabetes technology use and T1D health outcomes among Latinx adolescents. If found to be effective, the VPG curriculum can be adapted for other clinic settings in order to improve education and peer support for Latinx patients and families. Future studies may extend or adapt DREAM to other cohorts, including other age groups, geographic settings, or marginalized and historically excluded populations with T1D.

ELIGIBILITY:
Inclusion Criteria:

* Adolescents 13-17 years old and their caregivers
* Adolescent must have T1D of any duration, and be receiving diabetes care at UCSF, CHLA or UC Davis
* Self-identify as Latina/o/x or other variations such as Hispanic
* Preferred language of English or Spanish

Exclusion Criteria:

* Participants who have a medical, developmental, or psychiatric condition that would make peer group participation difficult
* Adolescents who are planning to transfer care to a different medical center within the next year, which would prevent assessment of longitudinal outcomes

Ages: 13 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 120 (Estimated)
Dates: Start 2024-10-11 (Actual); Primary Completion 2026-05-31 (Estimated); Study Completion 2026-05-31 (Estimated)

PRIMARY OUTCOMES:
Caregiver Survey | Baseline
  Captures personal and family background (e.g. gender, income)
Caregiver Phase 2 Intervention Survey - "Feedback Survey" | End of Study to (6-15 months)
  Assess various intervention components (e.g., frequency of virtual peer groups, in person events).
Caregiver In Person Event Evaluation | Throughout the study, up to 15 months
  Captures in the moment in person event feedback (e.g., improve experience and components).
Caregiver Online Group Evaluation | Throughout the study, up to 15 months
  Captures moment group feedback (e.g., improve experience and content).
Adolescent Survey | Baseline
  Captures diabetes technology, personal and family background (e.g., diabetes technology history, gender).
Adolescent Phase 2 Intervention Survey - "Feedback Survey" | End of Study (6-15 months)
  Assess various intervention components (e.g, frequency of virtual peer groups, in person events).
Adolescent In Person Event Evaluation | Throughout the study, up to 15 months
  Captures in the moment in person event feedback (e.g., improve experience and components).
Adolescent Online Group Evaluation | Throughout the study, up to 15 months
  Captures moment group feedback (e.g., improve experience and content).
Attendance at VPG and in-person events | Throughout the study, up to 15 months
  Attendance will be recorded for each in person and online events
Retention of enrolled patients | End of Study (6-15 months)
  Engagement of participants throughout study trajectory

SECONDARY OUTCOMES:
Caregiver Diabetes Distress Scale (DDS) | Baseline and End of Study (6-15 months)
  Measures parent-related distress, person distress, teen management distress, parent/teen relationship distress and healthcare distress, response options for each item were provided on a 5-point Likert scale, higher score indicated more distress.
Caregiver Diabetes Family Conflict Scale (DFCS) | Baseline and End of Study (6-15 months)
  Measures negative emotions around BGM, quality of life, and perceived parental burden from diabetes management; 3-point Likert scale, higher score indicating more conflict.
Caregiver Health Care Relationship (QHR) | Baseline and End of Study (6-15 months)
  Captures interactions with medical team, response options for each item were provided on a 5-point Likert scale in various formats.
Patient Health Utilization | Baseline, 3-months, 6-months, 9-months, End of Study 12 to 15-months
  Asks about any interval ED or hospital utilization over the prior 3 months
Adolescent Diabetes Distress Scale (DDS) | Baseline and End of Study (6-15 months)
  Measures diabetes emotional distress; response options for each item were provided on a 5-point Likert scale, higher score indicated more distress.
Adolescent Benefits and Burdens of CGM (BenCGM & BurCGM) | Baseline and End of Study (6-15 months)
  Measures benefits and burdens of continuous glucose monitoring in adolescents; 5-point Likert scale.
Adolescent Diabetes Family Conflict Scale, (DFCS) | Baseline and End of Study (6-15 months)
  Measures negative emotions around BGM, quality of life, and perceived parental burden from diabetes management, 3-point Likert scale, higher score indicating more conflict.
Adolescent Diabetes Strengths and Resilience Measure (DSTAR) | Baseline and End of Study (6-15 months)
  Captures adaptive aspects of adolescents' diabetes management (i.e., "strengths"), and is related to clinical outcomes, 5-point Likert scale.
Adolescent BenPump/Pod & BurPump/Pod | Baseline and End of Study (6-15 months)
  Measures benefits and burdens of pump/pods monitoring in adolescents, 5-point Likert scale.

OTHER OUTCOMES:
Socio-Demographic History | Baseline
  Self-reported demographic history (gender, age, race, household income, etc) will be collected.
Diabetes Technology Use | Baseline and End of Study (6-15 months)
  Diabetes technology use history self-reported and Electronic Medical Record (EMR) Abstraction
Number of participants completing rountine appointments | Baseline and End of Study (6-15 months)
  Electronic Medical Record (EMR) Abstraction
Hemoglobin A1c | Baseline and End of Study (6-15 months)
  Lab results

CONTACTS AND LOCATIONS:
Overall Officials: Jenise C Wong, MD, PhD, Principal Investigator — University of California, San Francisco
Locations (3):
- United States (3):
  - University of California, Davis, Davis, California
  - Children's Hospital Los Angeles, Los Angeles, California
  - University of California, San Francisco, San Francisco, California

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Hessler D, Fisher L, Polonsky W, Johnson N. Understanding the Areas and Correlates of Diabetes-Related Distress in Parents of Teens With Type 1 Diabetes. J Pediatr Psychol. 2016 Aug;41(7):750-8. doi: 10.1093/jpepsy/jsw002. Epub 2016 Feb 10. PMID 26869664
- [Background] Manning ML, Singh H, Stoner K, Habif S. The Development and Psychometric Validation of the Diabetes Impact and Device Satisfaction Scale for Individuals with Type 1 Diabetes. J Diabetes Sci Technol. 2020 Mar;14(2):309-317. doi: 10.1177/1932296819897976. Epub 2020 Feb 6. PMID 32028790
- [Background] Polonsky WH, Fisher L, Earles J, Dudl RJ, Lees J, Mullan J, Jackson RA. Assessing psychosocial distress in diabetes: development of the diabetes distress scale. Diabetes Care. 2005 Mar;28(3):626-31. doi: 10.2337/diacare.28.3.626. PMID 15735199
- [Background] Messer LH, Cook PF, Tanenbaum ML, Hanes S, Driscoll KA, Hood KK. CGM Benefits and Burdens: Two Brief Measures of Continuous Glucose Monitoring. J Diabetes Sci Technol. 2019 Nov;13(6):1135-1141. doi: 10.1177/1932296819832909. Epub 2019 Mar 10. PMID 30854886
- [Background] Hood KK, Butler DA, Anderson BJ, Laffel LM. Updated and revised Diabetes Family Conflict Scale. Diabetes Care. 2007 Jul;30(7):1764-9. doi: 10.2337/dc06-2358. Epub 2007 Mar 19. PMID 17372149
- [Background] Iturralde E, Hood KK, Weissberg-Benchell J, Anderson BJ, Hilliard ME. Assessing strengths of children with type 1 diabetes: Validation of the Diabetes Strengths and Resilience (DSTAR) measure for ages 9 to 13. Pediatr Diabetes. 2019 Nov;20(7):1007-1015. doi: 10.1111/pedi.12898. Epub 2019 Jul 29. PMID 31336011
- [Background] Hilliard ME, Iturralde E, Weissberg-Benchell J, Hood KK. The Diabetes Strengths and Resilience Measure for Adolescents With Type 1 Diabetes (DSTAR-Teen): Validation of a New, Brief Self-Report Measure. J Pediatr Psychol. 2017 Oct 1;42(9):995-1005. doi: 10.1093/jpepsy/jsx086. PMID 28549160